CLINICAL TRIAL: NCT07312734
Title: Study to Enable New Diagnostics for Pulmonary Microbes in People With CF (SEND-CF)
Brief Title: Study to Enable New Diagnostics for Pulmonary Microbes in People With CF
Acronym: SEND-CF
Status: Not yet recruiting | Type: Observational
Sponsor: Chris Goss (Other)
Collaborators: Cystic Fibrosis Foundation (Other); University of Pennsylvania (Other)
Responsible Party: Sponsor-Investigator, Chris Goss, Professor of Medicine and Pediatrics, University of Washington, Seattle Children's Hospital
Organization: Seattle Children's Hospital (Other)
Other Study IDs: SENDCF-OB-25
Record Dates: First submitted 2025-10-23; First posted 2025-12-31 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-10

CONDITIONS: Cystic Fibrosis (CF); New Diagnostics
Keywords: Cystic Fibrosis; CF; Breath collection; Specimen collection; Detection of pathogens; New diagnostics
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, plasma, buffy coat, urine, saliva, sputum, whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Sputum culture has been the best approach to detect harmful bacteria in the lungs of people with cystic fibrosis (CF). With the widespread use of new CF therapies (like Trikafta and Alyftrak), it is more difficult for people with CF to produce sputum even though they still have harmful bacteria in their lungs. The SEND-CF study is being done to see if there are other ways to detect harmful bacteria in the lungs.

DETAILED DESCRIPTION:
People with cystic fibrosis (CF) often get lung infections that can make their breathing worse and make their lungs weaker over time. Sputum culture is usually analyzed to find these infections. Currently, many people with CF are using CFTR modulators. These medicines help, but they also make it harder for people to cough up sputum. Even though people with CF are making less sputum, lung infections are still a problem. New ways are needed to check for infections without using sputum.

The SEND-CF study wants to gather health information and samples from people with CF in order to find new and better ways to spot harmful bacteria in the lungs. Participants, who typically are able to produce sputum who consent to participate will be asked to provide samples including sputum, saliva, serum, plasma, buffy coat, urine, and whole blood. Some participants will also provide breath samples for a sub-study.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 16 years of age on day of study visit
* Documentation of CF Diagnosis
* Able to expectorate sputum
* Percent predicted FEV1 ≥ 30%

Exclusion Criteria:

* History of solid organ transplantation
* History of active malignancy (or treatment for malignancy) in 12 months prior to the study visit
* Pregnant

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Study participants will be recruited at Cystic Fibrosis Foundation's Therapeutics Development Network study sites
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-08-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate alternative methods for the detection of microbial pathogens from the lungs of people with CF by comparing against the gold standard of sputum cultures. | Baseline Visit
  Specimens (including sputum, saliva, blood, urine, and breath (for the Owlstone Device Sub-Study)) will be collected at the Study Visit. These specimens will be stored at a biorepository and be made available to the research community to test and validate diagnostic assays for the detection of CF pathogens.

CONTACTS AND LOCATIONS:
Overall Officials: Gina Hong, MD, MHS, Principal Investigator — University of Pennsylvania
Locations (9):
- United States (9):
  - University of California San Diego, La Jolla, California
  - The Minnesota Cystic Fibrosis Center, Minneapolis, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Nationwide Children's Hospital, Columbus, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - University of Texas Southwestern, Dallas, Texas
  - Froedtert & Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No